CLINICAL TRIAL: NCT00695526
Title: Phase 3 Study of Cranberry on Lipid Profiles in Type 2 Diabetes
Brief Title: Effects of Cranberry Extractive on the Lipid Profiles in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Department of Medical Education and Research, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C06066
Record Dates: First submitted 2008-04-11; First posted 2008-06-12 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Type 2 Diabetes
Keywords: cranberry; total to HDL cholesterol ratio; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator)
  Interventions: Dietary Supplement: cranberry

INTERVENTIONS:
Dietary Supplement: cranberry — cranberry extractive in powder product (by Triarco Industries, Inc. NJ, USA) and encapsulated in dose of 500mg/capsule (by Topo digital tech co., Taiwan). By one capsule after each of three meals per day.

SUMMARY:
Cranberry, containing flavonoids, is effective on improvement of lipid profiles in non-diabetic subjects. The Hypothesis of is to assess the effect of cranberry on lipid profiles in type 2 diabetic patients using oral antidiabetic drugs.

DETAILED DESCRIPTION:
Hypercholesterolemia is a notorious risk factor for cardiovascular disease. It had been reported cranberry consumption increased nearly 8% of circulating high-density lipoprotein (HDL) cholesterol levels in non-diabetic subjects. Although characteristics of diabetic dyslipidemia are low HDL and high triglyceride, the benefits of concentrated powder of cranberry juice on lipid profiles were not evident in type 2 diabetic subjects with diet control alone. To the best of our knowledge, the effect of cranberry on lipid profiles in type 2 diabetic subjects using oral anti-diabetic drugs have never been studied, especially total to HDL cholesterol ratio which is important in predicting cardiovascular diseases in Asian and/or diabetic population. Furthermore, cranberry has anti-oxidative effect which is associated with reduction of oxidized low-density lipoprotein (ox-LDL) cholesterol in non-diabetes. Therefore, we conducted a placebo-controlled, double-blind, randomized study to assess the effect of cranberry on lipid profiles in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic subjects
* age between 50 and 75 years

Exclusion Criteria:

* glycosylated hemoglobin (HbA1c) less than 7% or more than 10%;
* triglyceride more than 4.5 mmol/L;
* current insulin treatment;
* change of the medications for anti-diabetes, hypertension, hyperlipidemia and anti-platelet in recent four weeks;
* abnormal renal function (serum creatinine > 177 μmol/L;
* abnormal liver function test results (more than two-fold upper limit of normal range);
* severe systemic disease such as immune disorder, cancer, acute or chronic inflammation disease;
* smoking in recent 1 year;
* alcoholism (more than two drinks daily);
* using steroid or drugs with unknown components;
* pregnancy or breast-feeding.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
the change of total to HDL cholesterol ratio | 12 weeks

SECONDARY OUTCOMES:
the change of lipid profiles (LDL, total cholesterol, HDL and triglyceride) | 12 weeks
the change of ox-LDL | 12 weeks
the change of fasting plasma glucose | 12 weeks
the change of HbA1c | 12 weeks
the change of CRP | 12 weeks
the change of UAE | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: I Te Lee, MD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- outpatient clinic of the Division of Endocrinology and Metabolism in Taichung Veterans General Hospital, Taichung, Taiwan